CLINICAL TRIAL: NCT00743236
Title: A Phase III Multi-Institutional Randomized Clinical Trial: Effect of Type of Ischemia - Warm vs Cold During Partial Nephrectomy - on Renal Function
Brief Title: Warm Ischemia or Cold Ischemia During Surgery in Treating Patients With Stage I Kidney Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCCWFU-89108; CDR0000612519 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-01120 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Kidney Cancer; Long-term Effects Secondary to Cancer Therapy in Adults; Perioperative/Postoperative Complications; Urinary Complications
Keywords: perioperative/postoperative complications; urinary complications; long-term effects secondary to cancer therapy in adults; stage I renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Postoperative Complications; Carcinoma, Renal Cell | interventions — Cold Ischemia; Warm Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients undergo warm ischemia followed by partial nephrectomy.
  Interventions: Procedure: warm ischemia procedure
- Arm II (Experimental): Patients undergo cold ischemia followed by partial nephrectomy.
  Interventions: Procedure: cold ischemia procedure

INTERVENTIONS:
Procedure: cold ischemia procedure — Cold ischemia followed by partial nephrectomy
  Arms: Arm II
Procedure: warm ischemia procedure — Warm ischemia followed by partial nephrectomy
  Arms: Arm I

SUMMARY:
RATIONALE: Warm ischemia is the clamping of blood vessels without cooling the kidney. Cold ischemia is the clamping of blood vessels with kidney cooling. It is not yet known whether warm ischemia is more effective than cold ischemia in patients undergoing surgery for stage I kidney cancer.

PURPOSE: This randomized phase III trial is studying warm ischemia to see how well it works compared with cold ischemia during surgery in treating patients with stage I kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of warm ischemia during partial nephrectomy on long-term renal function in patients with solitary stage I renal cortical tumor and normal contralateral kidney.

Secondary

* Determine to what degree the contralateral kidney compensates for the damage inflicted on the operated kidney during surgery.
* Determine the 1-year disease-specific and overall survival of these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo warm ischemia followed by partial nephrectomy.
* Arm II: Patients undergo cold ischemia followed by partial nephrectomy. Blood and urine samples are collected periodically after nephrectomy to assess renal function.

Patients are followed at 1, 3, 6, 9 , and 12 months after nephrectomy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solitary renal cortical tumor

  * Tumor size ≤ 4 cm
* Candidate for open partial nephrectomy

  * Expected ischemia time < 45 minutes
* Normal renal function, defined as glomerular filtration rate (GFR) > 60 mL/min
* No evidence of distant metastasis
* No evidence of local invasion of adjacent structures, including the adrenal gland
* No evidence of tumor extension into the renal venous system
* No evidence of ureteral obstruction on MAG-3 renal scan
* No family history of renal cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0
* Life expectancy > 5 years
* No prior malignancy, except for non-melanomatous skin cancer

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Creatinine clearance at 1 year | at 1 year after nephrectomy.
Estimated glomerular filtration rate (GFR) | at 1 year after nephrectomy.

SECONDARY OUTCOMES:
Evidence of local or metastatic recurrence | at 1 year after nephrectomy.
Cancer-specific survival | at 1 year after nephrectomy.
Overall survival | at 1 year after nephrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Pettus, MD, Study Chair — Wake Forest University Health Sciences
Locations (8):
- United States (8):
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No